CLINICAL TRIAL: NCT03958825
Title: Randomized Clinical Trial of Open Versus Laparoscopic Left Hepatic Sectionectomy in Treatment of Hepatolithiasis Within an Enhanced Recovery After Surgery Programme
Brief Title: Open Versus Laparoscopic Left Hepatic Sectionectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, hui hou, general surgery, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 520
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Hepatolithiasis; Laparoscopic Liver Resection; Open Liver Resection; Enhanced Recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open left hepatic sectionectomy (Active Comparator): patients undergoing open left hepatic sectionectomy within an enhanced recovery after surgery programme
  Interventions: Procedure: open left hepatic sectionectomy
- laparoscopic hepatic sectionectomy (Experimental): patients undergoing a laparoscopic left hepatic sectionectomy within an enhanced recovery after surgery programme
  Interventions: Procedure: laparoscopic hepatic sectionectomy

INTERVENTIONS:
Procedure: laparoscopic hepatic sectionectomy — patients undergoing a laparoscopic left hepatic sectionectomy within an enhanced recovery after surgery programme
  Other Names: open left hepatic sectionectomy
  Arms: laparoscopic hepatic sectionectomy
Procedure: open left hepatic sectionectomy — patients undergoing open left hepatic sectionectomy within an enhanced recovery after surgery programme
  Arms: open left hepatic sectionectomy

SUMMARY:
Laparoscopic left sectionectomy has been associated with shorter hospital stay and reduced overall morbidity compared with open left sectionectomy. Strong evidence has not, however, been provided.

DETAILED DESCRIPTION:
The application of laparoscopic technology to liver surgery has been developing rapidly, yet very few studies have been conducted to compare the outcomes between open and laparoscopic liver resections. So little is known about their advantages and disadvantages. The aim of this prospective randomized study is to compare the outcomes between laparoscopic and open liver resection in treatment of hepatolithiasis within the left lobes within an enhanced recovery after surgery programme.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for undergoing both laparoscopic left sectionectomy as well as open left sectionectomy of the liver
* Able to understand the nature of the study and what will be required of them
* Men and non-pregnant,non-lactating women between age 18-80
* BMI between 18-35
* Patients with ASA I-II-III

Exclusion Criteria:

* Inability to give written informed consent
* Patients undergoing liver resection other than left lateral hepatic sectionectomy
* Patients with ASA IV-V Underlying liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2022-12-26 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospital duration after operation (days) | up to 30 days after liver resection
  the length of hospital stay

SECONDARY OUTCOMES:
Readmission percentage | up to 30 days after liver resection
  Readmission percentage during one year follow-up
Total morbidity | up to 1 year after liver resection
  According to The Clavien-Dindo Classification, https://www.assessurgery.com/clavien-dindo-classification/
Composite endpoint of liver surgery specific morbidity | up to 1 year after liver resection
  Parameter composed of a combination of procedure-specific complications and considered as a single, dichotomous outcome: operative mortality, intra-abdominal haemorrhage, ascites, bile leakage, intra-abdominal abscess and postresectional liver failure. These components, which are all specific to liver surgery and have substantial clinical relevance, reflect Dindo grade 3-5 complications. A composite score of 1 (=failure) will reflect the occurrence of at least one of the above liver specific complications, consequently a score of 0 (=success) will be assigned if none occur.
Hospital and societal costs | up to 1 year after liver resection
  The economic evaluation will include a cost-utility analysis from a Dutch societal perspective. The incremental costs per Quality Adjusted Life Year (QALY) gained will be based on utility scores from the EQ-5D. All hospital expenses (direct and indirect) related to both interventions will be monitored. In addition, a cost questionnaire offered at the regular follow-up consultation (3, 6 and 12 months) will help us to assess the societal and individual costs outside health care relating to patients' absence, impaired mobility, work or normal daily activities.
Incidence of incisional hernias | up to 1 year after liver resection
  To assess the incidence of incisional hernias in laparoscopic and open left lateral hepatic sectionectomy patients will be contacted at a mean time of 1 year after resection to receive an ultrasound to diagnose incisional hernia.
Change of serum glutamic oxalacetic transaminase | up to 7 days after liver resection
  Change of serum glutamic oxalacetic transaminase after liver resection.These values will be recorded preoperative, and postoperative day-1,3,5,7.
Change of serum glutamic-pyruvic transaminase | up to 7 days after liver resection
  Change of serum glutamic-pyruvic transaminase after liver resection.These values will be recorded preoperative, and postoperative day-1,3,5,7.
Mortality rates | up to 30 days after liver resection
  the rate of postoperative death
Operation time(min) | intraoperative
  the during of operation
Blood loss(ml) | up to 30 days after liver resection
  the volume of blood loss
Blood transfusion (times and units) | intraoperative
  intraoperative blood transfusion
C-reactive protein (mg/mL) | up to 5 days after liver resection
  C-reactive protein levels on preoperative and postoperative day-1,3,5

CONTACTS AND LOCATIONS:
Overall Officials: hui hou, master, Study Chair — Second Affiliated Hospital of Anhui Medical University
Locations (1):
- The second hospital of Anhui Medical University,, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan SB, Wu CL, Zhou DC, Xiong QR, Geng XP, Hou H. Total laparoscopic partial hepatectomy versus open partial hepatectomy for primary left-sided hepatolithiasis: study protocol for a randomized controlled trial. Trials. 2024 Feb 22;25(1):137. doi: 10.1186/s13063-023-07476-w. PMID 38383461